CLINICAL TRIAL: NCT03065660
Title: A Randomised Placebo-controlled Trial of Mifepristone and Misoprostol Versus Misoprostol Alone in the Medical Management of Missed Miscarriage
Brief Title: Mifepristone and Misoprostol Versus Misoprostol Alone in the Medical Management of Missed Miscarriage
Acronym: MifeMiso
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Birmingham Women's NHS Foundation Trust (Other Government); Royal Infirmary of Edinburgh (Other); Royal Victoria Infirmary (Other); City Hospitals Sunderland NHS Foundation Trust (Other); Liverpool Women's NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); Barts & The London NHS Trust (Other); Queen's Medical Center (Other); Heart of England NHS Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); St Mary's Hospital, London (Other); University College London Hospitals (Other); University Hospital Southampton NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); University of Edinburgh (Other); University of Nottingham (Other); Queen Mary University of London (Other); University of Warwick (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RG_16-076; 15/160/02 (Other Grant/Funding Number: NIHR HTA); 2016-005097-35 (EudraCT Number)
Record Dates: First submitted 2017-02-10; First posted 2017-02-28 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Missed Miscarriage
Keywords: Missed miscarriage; Mifepristone; Misoprostol; Medical management
MeSH Terms: conditions — Abortion, Incomplete | interventions — Mifepristone

STUDY DESIGN:
Intervention Model Description: A randomised, parallel group, double-blind, placebo-controlled multicentre study, with health economic and mixed-methods evaluation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, investigators, research midwives/nurses and other attending clinicians will remain blind to the trial drug allocation throughout the duration of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mifepristone (Active Comparator): A single dose of oral mifepristone 200mg, followed by a single dose of vaginal, oral or sublingual misoprostol 800mcg 2 days later
  Interventions: Drug: Mifepristone, Oral, 200 Mg
- Placebo (Placebo Comparator): Oral placebo tablet followed by a single dose of vaginal, oral or sublingual misoprostol 800mcg 2 days later.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Mifepristone, Oral, 200 Mg — The Investigational Medicinal Product (IMP) is a single dose of 200mg mifepristone to be taken orally after confirmation of missed miscarriage by pelvic ultrasound scan.
  Other Names: Mifegyne
  Arms: Mifepristone
Drug: Placebo Oral Tablet — The placebo will be an oral tablet in the same form as the IMP, and identical in appearance.
  Arms: Placebo

SUMMARY:
Miscarriage is the most common complication of pregnancy. As many as 15-25% of pregnancies end in miscarriage, and the number of miscarriages in England is estimated to be approximately 125,000 per year. Miscarriage often brings not only physical pain, bleeding and risks of infection, but also psychological impacts on women and their families. This study will focus on women whose pregnancy sac remains inside the womb (known as a missed miscarriage) and opt for medical management of their miscarriage up to 13+6 weeks of pregnancy. NICE currently recommends that a drug called misoprostol (a vaginal pessary or oral tablet that makes the womb contract) should be used in the medical treatment of miscarriage. However, there is evidence to suggest that combining this drug with mifepristone (an oral tablet that reduces pregnancy hormones) may be more effective in treating miscarriage. Therefore, to test this in a clinical trial, participants will be allocated at random to receive either mifepristone followed by misoprostol, or a dummy drug (placebo) followed by misoprostol. Neither the participants nor the researchers will know what allocation is decided, which is necessary to test the treatments fairly. The main outcome of interest will be whether miscarriage is complete within 7 days of randomisation. If miscarriage is not complete then further treatment (more tablets or surgery) will be offered. A number of other key outcomes, such as the need for an operation, will also be assessed. We will also study the views and experience of the participants regarding the tablet treatment.

We anticipate that 710 women will be required to take part in the study to answer this question with confidence. We estimate that we would be able to recruit this many women in two years.

DETAILED DESCRIPTION:
Aim: To investigate the clinical and cost-effectiveness of MifeMiso combination (mifepristone and misoprostol) versus misoprostol alone in the management of missed miscarriage.

Primary clinical objective: To test the hypothesis that treatment with mifepristone plus misoprostol is superior to misoprostol alone for the resolution of miscarriage within 7 days in women diagnosed with missed miscarriage by pelvic ultrasound scan in the first 13+6 weeks of pregnancy.

Key secondary objective:To test the hypothesis that the addition of mifepristone reduces the need for surgical intervention to resolve the miscarriage.

Other secondary objectives:

1. To evaluate if the addition of mifepristone reduces the need for further doses of misoprostol.
2. To evaluate if the addition of mifepristone improves other clinical outcomes including surgical intervention up to and including 7 days post-randomisation and after 7 days post-randomisation, duration of bleeding, infection, negative pregnancy test at 21 days post-randomisation, time from randomisation to discharge from EPU care, side effects and complications.
3. To evaluate if the addition of mifepristone improves patient satisfaction
4. To assess the cost-effectiveness of the combination of mifepristone and misoprostol in the medical management of missed miscarriage.

Economic objectives: To assess the cost-effectiveness of the combination of mifepristone and misoprostol in the medical management of missed miscarriage based on an outcome of additional cost per additional successfully managed miscarriage and additional cost per additional quality-adjusted life-year (QALY). Using a model-based economic evaluation we will further explore the cost-effectiveness of the medical management of missed miscarriage, as explored in the proposed trial, with alternative management strategies, such as surgical and expectant, based on available secondary sources.

Mixed-method evaluation objectives: To explore the satisfaction of patients who complete the trial protocol. The results of the satisfaction survey (CSQ-8) will act as a sampling frame to conduct semi-structured interviews to further investigate patient experiences and satisfaction with medical management of missed miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with missed miscarriage by pelvic ultrasound scan in the first 13+6 weeks of pregnancy that choose to have medical management of miscarriage.
* Age 16 years and over
* Willing and able to give informed consent.

Exclusion Criteria:

* Women opting for alternative methods of miscarriage management (expectant or surgical)
* Diagnosis of incomplete miscarriage.
* Life threatening bleeding.
* Contraindications to mifepristone or misoprostol use for example chronic adrenal failure, known hypersensitivity to either drug, haemorrhagic disorders and anticoagulant therapy, prosthetic heart valve or history of endocarditis, existing cardiovascular disease, severe asthma uncontrolled by therapy or inherited porphyria.
* Participation in any other blinded, placebo-controlled trials of investigational medicinal products in pregnancy.
* Previous participation in the MifeMiso trial
* Woman not able to attend for day 6-7 ultrasound scan

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Failure to spontaneously pass the gestational sac within 7 days after randomisation | Within 7 days after randomisation
  To test the hypothesis that treatment with mifepristone plus misoprostol is superior to misoprostol alone for the resolution of miscarriage within 7 days in women diagnosed with missed miscarriage by pelvic ultrasound scan in the first 13+6 weeks of pregnancy.

SECONDARY OUTCOMES:
Surgical intervention to resolve the miscarriage (collected up to discharge from EPU care) | From randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Surgical intervention to resolve the miscarriage
Surgical intervention to resolve the miscarriage up to and including day 7 post-randomisation | From randomisation until day 7 post-randomisation
  Surgical intervention to resolve the miscarriage
Surgical intervention to resolve the miscarriage after day 7 post-randomisation to discharge from EPU care | From day 8 post-randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Surgical intervention to resolve the miscarriage
Need for further doses of misoprostol up to day 7 post-randomisation | After initial 800mcg dose of misoprostol at day 2 until day 7 post-randomisation
  Need for further doses of misoprostol up to day 7 post-randomisation
Need for further doses of misoprostol up to discharge from EPU care | After initial 800mcg dose of misoprostol at day 2 until discharge from EPU care; assessed up to approximately 8 weeks
  Need for further doses of misoprostol up to discharge from EPU care
Overall patient satisfaction score (measured using the CSQ-8 questionnaire and collected upon discharge from EPU care). | Within 6 weeks of discharge from EPU care
  Overall patient satisfaction score (measured using the CSQ-8 questionnaire and collected upon discharge from EPU care).
Patient quality of life (Index value and overall health status measured using the EQ-5D-5L questionnaire | Completion on date of randomisation, day 6-7 post-randomisation or day of follow-up USS if different to day 6-7 and day 21 +/- 2 days post-randomisation. Completion of all patient quality of life assessments up to approximately 8 weeks post-randomisation
  Patient quality of life (Index value and overall health status measured using the EQ-5D-5L questionnaire and collected on date of randomisation, day 6-7 post-randomisation or day of follow-up USS if different to day 6-7 and day 21 +/- 2 days post-randomisation. If a woman obtains an initial positive pregnancy test result at day 21 +/- 2 days post-randomisation then a further EQ-5D-5L questionnaire is collected upon discharge from EPU care).
Duration of bleeding reported by woman (days). (collected up to discharge from EPU care) | From randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Duration of bleeding reported by woman (days). (collected up to discharge from EPU care)
Diagnosis of infection associated with miscarriage requiring outpatient antibiotic treatment (collected up to discharge from EPU care) | From randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Diagnosis of infection associated with miscarriage requiring outpatient antibiotic treatment (collected up to discharge from EPU care)
Diagnosis of infection associated with miscarriage requiring inpatient antibiotic treatment (collected up to discharge from EPU care) | From randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Diagnosis of infection associated with miscarriage requiring inpatient antibiotic treatment (collected up to discharge from EPU care)
Negative pregnancy test result 21 days (± 2 days) after randomisation. | 21 days (± 2 days) after randomisation.
  Negative pregnancy test result 21 days (± 2 days) after randomisation.
Time from randomisation to discharge from EPU care (described using summary statistics only) | Time from randomisation to discharge from EPU care; assessed up to approximately 8 weeks
  Time from randomisation to discharge from EPU care.
Blood transfusion required (collected up to discharge from EPU care) | From randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Blood transfusion required (collected up to discharge from EPU care)
Side effects (collected up to discharge from EPU care) | From randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Side effects (collected up to discharge from EPU care)
Death (collected up to discharge from EPU care) | From randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Death (collected up to discharge from EPU care)
Any serious complications (collected up to discharge from EPU care) | From randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Any serious complications (collected up to discharge from EPU care)

OTHER OUTCOMES:
Outpatient or emergency visits | From randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Number of outpatient or emergency visits
Inpatient admissions (nights in hospital) | From randomisation until discharge from EPU care; assessed up to approximately 8 weeks
  Number of inpatient admissions (nights in hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Arri Coomarasamy, Principal Investigator — University of Birmingham
Locations (28):
- United Kingdom (28):
  - Birmingham Heartlands Hospital, Birmingham
  - Birmingham Women's Hospital, Birmingham
  - Southmead Hospital, Bristol
  - St Michael's Hospital, Bristol
  - Burnley General Hospital, Burnley
  - University Hospital Coventry, Coventry
  - Royal Infirmary of Edinburgh, Edinburgh
  - Epsom Hospital, Epsom
  - St Helier Hospital, Epsom
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Liverpool Women's Hospital, Liverpool
  - Chelsea and Westminster Hospital, London
  - Kings College Hospital, London
  - Newham University Hospital, London
  - Royal London Hospital, London
  - St Thomas' Hospital, London
  - University College Hospital London, London
  - West Middlesex Hospital, London
  - Whipps Cross University Hospital, London
  - Royal Victoria Infirmary, Newcastle
  - Queen's Medical Centre, Nottingham
  - Queen Alexandra Hospital, Portsmouth
  - Princess Anne Hospital, Southampton
  - Sunderland Royal Hospital, Sunderland
  - Princess of Wales Hospital, Swansea
  - Singleton Hospital, Swansea
  - Princess Royal Hospital, Telford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial website — https://www.birmingham.ac.uk/mifemiso